CLINICAL TRIAL: NCT04582201
Title: A Phase 1 Study of agenT-797 to Treat Moderate to Severe Acute Respiratory Syndrome in COVID-19 Patients
Brief Title: A Clinical Trial to Evaluate the Safety of agenT-797 in COVID-19 Participants With ARDS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MiNK Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-1300-01
Record Dates: First submitted 2020-10-06; First posted 2020-10-09 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Respiratory Distress Syndrome, Adult
Keywords: SARS-CoV-2
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dosage and Cohorts (Experimental): Cohort 1: 100 × 10^6 iNKT cells; Cohort 2: 300 × 10^6 iNKT cells; Cohort 3: 1000 × 10^6 iNKT cells
  Dosage Frequency and Mode of Administration: agenT-797 will be administered to hospitalized participants as a single intravenous infusion.
  Interventions: Drug: agenT-797

INTERVENTIONS:
Drug: agenT-797 — agenT-797 is an off-the-shelf cell therapy consisting of ≥ 95% allogeneic human unmodified iNKT cells isolated from 1 healthy donor mononuclear cell apheresis unit and expanded ex vivo.

SUMMARY:
A Phase 1 study of agenT-797 to treat moderate to severe acute respiratory syndrome in Coronavirus disease 2019 (COVID-19) participants.

DETAILED DESCRIPTION:
This is a Phase 1 study to evaluate the safety and efficacy of agenT-797, an unmodified, allogeneic invariant natural killer T cells (iNKT) therapy, in participants with COVID-19, requiring mechanical ventilation, and with moderate to severe acute respiratory distress syndrome (ARDS) as determined by the Berlin definition.

The study will be conducted in 2 parts. Part 1 will employ a standard 3+3 dose escalation design of agenT-797. All participants will receive a single infusion of agenT-797. Participants will also receive other treatments and supportive care per discretion of the principal investigator. Once the maximum tolerated dose of agenT-797 has been cleared in Part 1, Part 2 of the study will be opened and enroll eligible participants in the Expansion Cohort.

A safety monitoring committee will be established to assess safety and decide on escalation to next cohort and expansion dose, as well as any protocol modification to include less severe cases.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily agree to participate and ability to provide informed consent or have duly appointed health care proxy with the authority to consent.
* Confirmed diagnosis of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection by polymerase chain reaction test or equivalent approved test.
* Inpatient hospitalization.
* Evidence of SARS-CoV-2 infection with the diagnosis of moderate to severe ARDS per Berlin definition, no more than 2 weeks prior to study enrollment.
* Participants, or duly appointed health care proxy with the authority to consent, must consent to placement of a central venous access line for the administration of agenT-797.

Exclusion Criteria:

* Currently participating and receiving study therapy of an investigational agent that is not registered for any other indication. Note: Participants may receive the standard of care for SARS-CoV-2 infection as per institutional practices.
* Presence of comorbidities limiting expected survival of <1 month.
* Any comorbidity which in the opinion of the investigator may preclude/confound study required safety and efficacy assessments.
* Clinically significant cardiomyopathy.
* Receipt of non-oncology vaccines containing live virus for prevention of infectious diseases within 4 weeks prior to first dose of study treatment.
* Known hypersensitivity to natural killer cells or their preservation solution.
* Active systemic bacterial or fungal infection or viral co-infection.
* Legally incapacitated or has limited legal capacity.
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2023-04-23 (Actual); Study Completion 2023-04-23 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events | Baseline through Month 6
Number of Participants with Dose-limiting Toxicities | Baseline through Month 6

SECONDARY OUTCOMES:
Time to Extubation | Up to Day 30
Change from Baseline in C-reactive Protein (CRP) | Baseline through Day 30 (every 12 hours, as feasible)
  CRP levels will be used to assess cytokine release syndrome.
All-cause Mortality | Day 30 and Month 6
Decay in Quantitative Viral Burden from Upper and Lower Respiratory Tract Samples | Day 30
Change from Baseline at Day 30 in Number of Allogeneic iNKT Cells | Baseline, Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — MiNK Therapeutics
Locations (3):
- United States (3):
  - Saint John's Cancer Institute, Santa Monica, California
  - Norton Cancer Institute, St. Matthews Campus, Louisville, Kentucky
  - Weill Cornell Medicine New York Presbyterian, New York, New York